CLINICAL TRIAL: NCT06391021
Title: Comparison Between Combined Scoring of Bethesda Cytology and TIRADS Ultrasound With Post- Operative Histopathology in Thyroid Nodule
Brief Title: Comparison Between Combined Scoring of Bethesda Cytology and TIRADS Ultrasound With Histopathology in Thyroid Nodule
Acronym: TIRADS
Status: Completed | Type: Observational
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Anupama Marasini, Intern Doctor, Department of Ear, Nose and Throat Head and Neck Surgery, Tribhuvan University, Nepal
Other Study IDs: 628
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Nodule
Keywords: FNAC; TIRADS; Bethesda; Histopathology
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A thyroid nodule is a discrete lesion within the thyroid gland that is radiologically distinct from the surrounding thyroid parenchyma. Most thyroid nodules are benign, with only 10% to 15% harboring cancer. This is a prospective study conducted at the department of Ear, Nose and Throat - Head and Neck Surgery (ENT-HNS) of Shree Birendra Hospital , a tertiary heath care centre of Nepal. Individuals visiting ENT-HNS outpatient department with thyroid nodules had undergone Ultrasonography (USG) of neck followed by Fine-Needle Aspiration Cytology (FNAC) from the thyroid nodules. USG was reported by Thyroid Imaging Reporting and Data System(TIRADS) and FNAC by Bethesda system. Thereafter patients were planned either for surgery either total thyroidectomy or hemithyroidectomy. Post operative histopathology was correlated with preoperative FNAC and USG reports.

DETAILED DESCRIPTION:
The main objective of this prospective cohort study is to know the correlation between pre- operative Bethesda with post- operative histopathology , pre - operative TIRADS with post operative Histopathology and comparison of combined scoring of Bethesda and TIRADS with histopathology report. It is of utmost importance to deep dive into thyroid nodules workup to detect malignant nodules, as the management aspect of benign and malignant nodules has a vast difference. Thyroid ultrasonography is useful for risk stratification of nodules, and American College of Radiology Thyroid Imaging Reporting and Data System (ACR TI-RADS) classification provides recommendations for fine-needle aspiration cytology (FNAC) based on objective ultrasonography features of these nodules. To maintain uniformity in reporting system FNA sample are categorized according to the Bethesda system. Total 42 participants who met the inclusion criteria were included in the study. Statistical Analysis was done using Statistical Package for the Social Science (SPSS) version 25. Analysis was done in the form of percentage and proportion and represented as table wherever necessary. Spearman's correlation coefficient was used to evaluate the correlation between Bethesda and TIRADS. Bethesda and histopathology and TIRADS and Bethesda system. The P value was set at < 0.05 for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients presenting to Ear Nose and Throat, Head and Neck Surgery Department with thyroid nodules undergoing hemithyroidectomy or total thyroidectomy within the study period

Exclusion Criteria:

* 1.Patients refusing to give consent for the study. 2.Patients with already known case of thyroid malignancies proven by histopathological reports.

Ages: 20 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the participants with thyroid nodules who met the inclusion criteria within the study period were enrolled in the study . Total 42 participants were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Correlation between Bethesda and TIRADS system | 6 months
  Correlation between Bethesda and TIRADS system in terms of number of participants belonging to each category
Performance measure of Bethesda classification | 6 months
  Performance measure of Bethesda classification in terms of percentage
Performance measure of TIRADS classification | 6 months
  Performance measure of TIRADS classification in terms of percentage

SECONDARY OUTCOMES:
Sex-wise Distribution of thyroid nodule | 6 months
  Sex-wise Distribution of thyroid nodule in percentage
Percentage of participants as per TIRADS classification | 6 months
  Percentage of participants as per TIRADS classification
Number of participants as per histopathological examination | 6 months
  Number of participants as per histopathological examination
Number of participants as per Bethesda classification | 6 months
  Number of participants as per Bethesda classification
Types of surgical procedures performed in terms of percentage | 6 months
  Types of surgical procedures performed in terms of percentage

CONTACTS AND LOCATIONS:
Overall Officials: Reeba Karki, MS, Principal Investigator — Shree Birendra Hospital
Locations (1):
- Shree Birendra Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data to protect the privacy of the participants.

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967